CLINICAL TRIAL: NCT03545919
Title: Clinical Significance of Community-acquired Respiratory Virus Infection and Longitudinal Analysis of the Lung Microbiome in Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bin Cao, Doctor of Medicine, Capital Medical University
Other Study IDs: 2018-20-K15
Record Dates: First submitted 2018-05-13; First posted 2018-06-04 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Lung Transplant Infection; Lung Transplant Rejection
Keywords: respiratory viral infections; chronic lung allograft dysfunction; lung microbiome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the clinical significance of community-acquired respiratory virus (CARV) infection in patients with lung transplantation;Explore the lung microbiome dynamics within one year after lung transplantation;Find the relationship between lung microbiome and chronic lung allograft dysfunction(CLAD).

DETAILED DESCRIPTION:
Title:Clinical Significance of Community-acquired Respiratory Virus Infection and Longitudinal Analysis of the Lung Microbiome in Lung Transplantation.

Background:Infection affects the short-term prognosis of patients with lung transplantation and chronic lung allograft dysfunction(CLAD) limits their long-term survival.It is important to provide more theoretical support for early diagnosis and treatment of acute respiratory tract infection and CLAD in patients with lung transplantation.

Study Objectives:Evaluate the clinical significance of community-acquired respiratory virus (CARV) infection in patients with lung transplantation;Explore the lung microbiome dynamics within one year after lung transplantation;Find the relationship between lung microbiome and CLAD.

Study Design:A prospective and longitudinal study,following up the patients for 3 years.

Sample Size:100 cases. Study methods:CARV detection for respiratory specimens are performed during acute infection and routine re-testing in patients after lung transplantation,following up the patients who have positive findings to analyze the progression rates to lower respiratory tract infection,mortality rate within 90 days and risk factors associated with progression and death.For HRV/CoVs/HBoV detecting positive patients, consecutively collect respiratory specimens to quantitate viral load and combine virus serology to further confirm their pathogenicity on host.Complete a longitudinal 16S ribosomal RNA and metagenomics survey of the lung microbiome on respiratory samples collected from routine testing or re-testing（pre-operation,24 hours after the operation，day 3, day 7, week 2, week 3, month 1, month 3, month 6, month 9, month 12 , month 18, month 24, month 30, month 36) to explore the lung microbiome dynamics within one year after lung transplantation and find the relationship between lung microbiome and CLAD after 3 years follow-up.Besides,collect the peripheral blood of some patients for transcriptome and/or whole genome sequencing to screen for the host susceptibility genes.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with lung transplantation. 2.The patients who agree to participate in this study and sign informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with lung transplantation who meet the below inclusion criteria will be recruited in China-Japan Friendship Hospital in Beijing,China.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-05 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The progression rates from upper respiratory tract infection to lower respiratory tract infection within 40 days after diagnosis. | 40 days after diagnosis
  CARV detection for respiratory specimens are performed during acute infection and routine re-testing in patients after lung transplantation,following up the patients who have positive findings to analyze the progression rates to lower respiratory tract infection.
Mortality rate within 90 days after diagnosis of respiratory viral infections | 90 days after diagnosis of respiratory viral infections
  CARV detection for respiratory specimens are performed during acute infection and routine re-testing in patients after lung transplantation,following up the patients who have positive findings to analyze mortality rate within 90 days after diagnosis of respiratory viral infections
Explore the lung microbiome dynamics within one year after lung transplantation. | 1 year follow-up after lung transplantation
  Complete a longitudinal 16S ribosomal RNA and metagenomics survey of the lung microbiome on respiratory samples collected from routine testing or re-testing（pre-operation,24 hours after the operation，day 3, day 7, week 2, week 3, month 1, month 3, month 6, month 9, month 12)
Whether chronic lung allograft dysfunction occurs for individuals after 3 years follow-up after lung transplantation and find the relationship between lung microbiome and CLAD | 3 years follow-up after lung transplantation
  Complete a longitudinal 16S ribosomal RNA and metagenomics survey of the lung microbiome on respiratory samples collected from routine testing or re-testing（24 hours after the operation，month 3, month 6, month 9, month 12 , month 18, month 24, month 30, month 36)

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chambers DC, Yusen RD, Cherikh WS, Goldfarb SB, Kucheryavaya AY, Khusch K, Levvey BJ, Lund LH, Meiser B, Rossano JW, Stehlik J; International Society for Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: Thirty-fourth Adult Lung And Heart-Lung Transplantation Report-2017; Focus Theme: Allograft ischemic time. J Heart Lung Transplant. 2017 Oct;36(10):1047-1059. doi: 10.1016/j.healun.2017.07.016. Epub 2017 Jul 19. No abstract available. PMID 28784324
- [Result] Peghin M, Hirsch HH, Len O, Codina G, Berastegui C, Saez B, Sole J, Cabral E, Sole A, Zurbano F, Lopez-Medrano F, Roman A, Gavalda J. Epidemiology and Immediate Indirect Effects of Respiratory Viruses in Lung Transplant Recipients: A 5-Year Prospective Study. Am J Transplant. 2017 May;17(5):1304-1312. doi: 10.1111/ajt.14042. Epub 2016 Oct 14. PMID 27615811
- [Result] Bridevaux PO, Aubert JD, Soccal PM, Mazza-Stalder J, Berutto C, Rochat T, Turin L, Van Belle S, Nicod L, Meylan P, Wagner G, Kaiser L. Incidence and outcomes of respiratory viral infections in lung transplant recipients: a prospective study. Thorax. 2014 Jan;69(1):32-8. doi: 10.1136/thoraxjnl-2013-203581. Epub 2013 Sep 11. PMID 24025442
- [Result] Seo S, Gooley TA, Kuypers JM, Stednick Z, Jerome KR, Englund JA, Boeckh M. Human Metapneumovirus Infections Following Hematopoietic Cell Transplantation: Factors Associated With Disease Progression. Clin Infect Dis. 2016 Jul 15;63(2):178-85. doi: 10.1093/cid/ciw284. Epub 2016 May 3. PMID 27143659
- [Result] Bernasconi E, Pattaroni C, Koutsokera A, Pison C, Kessler R, Benden C, Soccal PM, Magnan A, Aubert JD, Marsland BJ, Nicod LP; SysCLAD Consortium. Airway Microbiota Determines Innate Cell Inflammatory or Tissue Remodeling Profiles in Lung Transplantation. Am J Respir Crit Care Med. 2016 Nov 15;194(10):1252-1263. doi: 10.1164/rccm.201512-2424OC. PMID 27248293
- [Result] Mouraux S, Bernasconi E, Pattaroni C, Koutsokera A, Aubert JD, Claustre J, Pison C, Royer PJ, Magnan A, Kessler R, Benden C, Soccal PM, Marsland BJ, Nicod LP; SysCLAD Consortium. Airway microbiota signals anabolic and catabolic remodeling in the transplanted lung. J Allergy Clin Immunol. 2018 Feb;141(2):718-729.e7. doi: 10.1016/j.jaci.2017.06.022. Epub 2017 Jul 18. PMID 28729000
- [Result] Willner DL, Hugenholtz P, Yerkovich ST, Tan ME, Daly JN, Lachner N, Hopkins PM, Chambers DC. Reestablishment of recipient-associated microbiota in the lung allograft is linked to reduced risk of bronchiolitis obliterans syndrome. Am J Respir Crit Care Med. 2013 Mar 15;187(6):640-7. doi: 10.1164/rccm.201209-1680OC. Epub 2013 Jan 17. PMID 23328523
- [Result] Borewicz K, Pragman AA, Kim HB, Hertz M, Wendt C, Isaacson RE. Longitudinal analysis of the lung microbiome in lung transplantation. FEMS Microbiol Lett. 2013 Feb;339(1):57-65. doi: 10.1111/1574-6968.12053. Epub 2012 Dec 20. PMID 23173619